CLINICAL TRIAL: NCT02345941
Title: Evaluating a Web-based Child Passenger Safety Program: Safety in Seconds 2.0
Brief Title: Safety in Seconds 2.0: An App to Increase Car Seat Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Andrea Gielen, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD069221-01A1
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Invervention (Experimental): The intervention group will get tailored information on the Parent Action Report and the Parent Portal about child safety seats and booster seats.
  Interventions: Other: Parent Action Report; Other: Parent Portal
- Control (Active Comparator): The control group will get tailored information in the Parent Action Report and the Parent Portal about smoke alarms.
  Interventions: Other: Parent Action Report; Other: Parent Portal

INTERVENTIONS:
Other: Parent Action Report — Parent Action Report will be displayed after the baseline assessment and contain educational safety messages.
Other: Parent Portal — Parents will have access to the Parent Portal, and they will be encouraged to visit it at any time.

SUMMARY:
This project will utilize the first web-based program to provide tailored injury prevention education. The existing Safety in Seconds program was adapted into a smartphone platform. Parents are recruited from and engage in the program in the clinical setting (PED or PTS). Parents download the app onto their smartphone which is used to ask the questions, collect a parent's responses, assess the parents' safety needs and give tailored directions for proper car sear use. The control group parents will also engage with the smartphone app and receive immediate feedback. However, they will receive tailored educational messages about smoke alarms. Parents will also have access to the online SIS v 2.0 Parent Portal which will have educational features (e.g., tips for keeping children content in their CSSs, links to helpful websites). The investigators will use emerging technology such as push notification and email to remind parents to visit the portal and have their child's car seat reassessed.

The investigators plan to conduct a cost benefit analysis of the program's expected financial benefit from the perspective of a third party payer of medical claims and an in-depth examination of program adoption and implementation using qualitative data collected from key informant interviews, direct observations of the clinic environments, and document review.

ELIGIBILITY:
Inclusion Criteria:

* Visiting the Pediatric Emergency Department (PED) at Johns Hopkins Hospital or Arkansas Children's Hospital
* Parent or guardian of child 4-7 years
* English speaking
* Have and Android or iPhone smartphone
* Drive with the child in a car at least once per week in a car that the parent owns, borrows or gets a ride round-trip
* Resident of Baltimore City, MD or Little Rock, AR and surrounding area.

Exclusion Criteria:

* PED has flagged case as suspected abuse
* Another household member is enrolled in the study
* In Arkansas, less than 18 years without parent present at the PED

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline self-reported car seat use at 6 months | 6 months
  Self-reported measures include the type of car seat used (rear-facing car seat, forward-facing car seat, booster seat, or seat belt), the location in car where it is used (front seat or backseat), frequency of use (some of the time or all of the time) and having the seat inspected by a car seat technician.

SECONDARY OUTCOMES:
Change from baseline self-reported smoke alarm use at 6 months | 6 months
  Self-reported measures include having a smoke alarm on every level of the home, having long-life battery alarms in the home, having a fire escape plan and practicing the fire escape plan.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Gielen, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Elise C Omaki, MHS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Johns Hopkins School of Public Health, Baltimore, Maryland

REFERENCES:
- [Derived] Gielen AC, Bishai DM, Omaki E, Shields WC, McDonald EM, Rizzutti NC, Case J, Stevens MW, Aitken ME. Results of an RCT in Two Pediatric Emergency Departments to Evaluate the Efficacy of an m-Health Educational App on Car Seat Use. Am J Prev Med. 2018 Jun;54(6):746-755. doi: 10.1016/j.amepre.2018.01.042. Epub 2018 Apr 12. PMID 29656914
- [Derived] Omaki E, Shields WC, McDonald E, Aitken ME, Bishai D, Case J, Gielen A. Evaluating a smartphone application to improve child passenger safety and fire safety knowledge and behaviour. Inj Prev. 2017 Feb;23(1):58. doi: 10.1136/injuryprev-2016-042161. Epub 2016 Sep 5. PMID 27597399